CLINICAL TRIAL: NCT03032107
Title: A Phase 1b Study Of Pembrolizumab In Combination With Trastuzumab-DM1 In Metastatic HER2-Positive Breast Cancer
Brief Title: A Study Of Pembrolizumab In Combination With Trastuzumab-DM1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-492
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Results first posted 2024-12-02 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Combine With Trastuzumab Emtansine (Experimental): * Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * Pembrolizumab will be administered prior to T-DM1 administration
  * Pembrolizumab will be given at a predetermine dose
  * T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * T-DM1 will be given at a predetermine dose
  Interventions: Drug: T-DM1; Drug: Pembrolizumab

INTERVENTIONS:
Drug: T-DM1 — -T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  Other Names: Trastuzumab emtansine
Drug: Pembrolizumab — -Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
  Other Names: Keytruda

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for metastatic breast cancer.

The interventions involved in this study are:

* Pembrolizumab
* Trastuzumab emtansine (also called T-DM1)

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved the combination of Pembrolizumab and T-DM1 for use in patients, including people with your type of cancer.

This study will determine what amount (or dose) of Pembrolizumab and of T-DM1 is safe for people to take and what effects, good or bad, this combination may have on participants and their disease.

The FDA has not approved Pembrolizumab for this specific disease but it has been approved in the United Sates for the treatment of other types of cancer.

The FDA has approved Trastuzumab emtansine (T-DM1) as a treatment option for this type of breast cancer

The combination of Pembrolizumab and T-DM1 is investigational. It is thought that together these drugs to help get the immune system to attack tumor cells and kill cancer cells that have the HER2 protein. However, it is not known if giving the two study drugs at the same time will have a better anti-cancer effect than giving each treatment on its own.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Either the primary tumor and/or the metastasis must have been tested for ER, PR and HER2. Patient must have HER2+ breast cancer per ASCO CAP guidelines 2013.
* Prior chemotherapy:

  * History of prior therapy with trastuzumab and a taxane, separately or in combination, is required.
  * Patients must have either received one line of prior therapy for metastatic breast cancer, or have developed a disease recurrence during or within 6 months after completing adjuvant therapy.
  * No prior treatment with T-DM1 is allowed.
  * Last dose of chemotherapy must be at least 21 days prior to registration.
* Prior biologic therapy:

  --Patients must have discontinued all biologic or investigational therapy at least 21 days before registration.
* Prior radiation therapy:

  * Patients may have received prior radiation therapy in either the metastatic or early-stage setting.
  * Radiation therapy must be completed at least 14 days prior to registration.
* In the dose de-escalation cohort: Subjects must have evaluable disease. In the expansion cohort: Subjects must have at least one lesion that is not within a previously radiated field that is measurable on computerized tomography (CT) or magnetic resonance imaging (MRI) scan per RECIST version 1.1. Bone lesions are not considered measurable by definition.
* Age is ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/μl
  * platelets ≥100,000/μl
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤1.5mg/dL (≤2.0 in patients with known Gilberts syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN. ≤5.0 × institutional ULN for patients with documented liver metastases.
  * albumin >2.5mg/dL
  * serum creatinine ≤1.5mg/dL or calculated GFR ≥60 mL/min
  * INR/PT ≤1.5 times ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT/PTT ≤1.5 times ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Participants enrolling in the dose expansion must have tissue that is amenable to biopsy and be willing to undergo a fresh tissue biopsy at baseline. Participants who undergo an attempted research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are not required to undergo a repeat biopsy in order to continue on protocol.
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason and because tratuzumab, a component of T-DM1, is known to be teratogenic, women of child-bearing potential and men of childbearing potential must agree to use adequate contraception starting with the first dose of study therapy, for the duration of study participation, and for an additional 120 days after the last dose of study medication. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the treating physician and principal investigator should be informed immediately.
  * While on the study, women should not breast-feed.
  * Subjects of childbearing potential are defined as those who have not been surgically sterilized and/or have had a menstrual period in the past year
* Female subject of child-bearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Patients on bisphosphonates may continue receiving bisphosphonate therapy during study treatment.
* Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by echocardiogram or MUGA documented within 28 days prior to first dose of study drug.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The subject has received another investigational agent within 21 days of the first dose of study drug.
* The subject has received prior pembrolizumab or any other anti-PD-1 , anti-PD-L1, or anti-PD-L2 therapy, or has participated in any prior studies involving pembrolizumab.
* Pre-existing neuropathy greater than or equal to grade 2.
* Hypersensitivity to pembrolizumab or T-DM1 or any of their excipients.
* The subject has any history or evidence of active, non-infectious pneumonitis or interstitial lung disease.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least one month prior to trial therapy initiation, are neurologically stable with an absence of new neurological symptoms for at least 4 weeks prior to study entry, and have recovered from effects of radiotherapy or surgery. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before the first study drug. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician.
* Known carcinomatous meningitis.
* The subject has an uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure (New York Heart Association Class III or IV; see Appendix B), active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, chronic liver or renal disease, or severe malnutrition.
* Concurrent use of potent CYP3A4 inhibitors (see Appendix C), such as ketoconazole and erythromycin, should be avoided during the study treatment with T-DM1.
* Active infection requiring intravenous antibiotics at cycle 1 day 1.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the study sponsor to determine eligibility.
* The subject has a medical condition that requires chronic systemic steroid therapy or any other form of immunosuppressive medication including disease modifiying agents, or has required such therapy in the last 2 years. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* The subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.
* The participant is positive for Hepatitis B surface antigen, or Hepatitis C RNA.
* Known HIV-positive participants. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections with bone marrow suppressive therapy, i.e. nab-paclitaxel. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* The subject has received a live vaccine within 28 days of planned start of study therapy. Note: seasonal influenza vaccines for infection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (i.e. Flu-Mist ®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waks AG, Keenan TE, Li T, Tayob N, Wulf GM, Richardson ET 3rd, Attaya V, Anderson L, Mittendorf EA, Overmoyer B, Winer EP, Krop IE, Agudo J, Van Allen EM, Tolaney SM. Phase Ib study of pembrolizumab in combination with trastuzumab emtansine for metastatic HER2-positive breast cancer. J Immunother Cancer. 2022 Oct;10(10):e005119. doi: 10.1136/jitc-2022-005119. PMID 36252998

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab Combine With Trastuzumab Emtansine: * All patients were treated at dose level 1: 200mg Pembro + 3.6mg/kg T-DM1
  * Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * Pembrolizumab will be administered prior to T-DM1 administration
  * Pembrolizumab will be given at a predetermine dose
  * T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * T-DM1 will be given at a predetermine dose
  T-DM1: -T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  Pembrolizumab: -Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
Period: Dose De-escalation (Dose-finding)
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Started | 6
Completed | 6 (All patients in this period were treated with dose level 1: 200mg Pembro + 3.6mg/kg T-DM1. Dose level 1 will be used in the expansion period.)
Not Completed | 0
Period: Recommended Phase 2 Dose Expansion
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Started | 14 (It is the expansion cohort. All patients in this period received dose level 1: 200mg Pembro + 3.6mg/kg T-DM1)
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab Combine With Trastuzumab Emtansine: * All patients received 200mg Pembro + 3.6mg/kg T-DM1
  * Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * Pembrolizumab will be administered prior to T-DM1 administration
  * Pembrolizumab will be given at a predetermine dose
  * T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * T-DM1 will be given at a predetermine dose
  T-DM1: -T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  Pembrolizumab: -Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 54 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
ECOG at baselin [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). This is a numbering scale of 0 to 5. The higher the number, the worse the performance status. Zero (0) refers to being full active. 5 is dead.
  Participants
    0 | 14
    1 | 5
    2 | 1
ER/PR status at initial diagnosis [Count of Participants; unit: Participants] — ER: Estrogen receptors PR: progesterone receptors
  Participants
    ER and/or PR positive | 14
    ER and PR negative | 6
Disease-free interval [Count of Participants; unit: Participants] — time from primary diagnosis to metastatic diagnosis
  Participants
    ≤2 years | 5
    >2 years | 6
    Dates missing | 4
    De novo (metastatic disease at primary diagnosis) | 5
Lines of chemotherapy for metastatic disease [Median (Full Range); unit: Line] | 1 [0 to 2]
Disease sites at trial enrollment - Lymph node [Count of Participants; unit: Participants] | 13
Disease sites at trial enrollment - Breast/chest wall [Count of Participants; unit: Participants] | 10
Disease sites at trial enrollment - Lung/pleura [Count of Participants; unit: Participants] | 9
Disease sites at trial enrollment - Bone [Count of Participants; unit: Participants] | 9
Disease sites at trial enrollment - Liver [Count of Participants; unit: Participants] | 4
Disease sites at trial enrollment - Other soft tissue [Count of Participants; unit: Participants] | 3
Disease sites at trial enrollment - Central nervous system [Count of Participants; unit: Participants] | 1
Prior therapy in any setting - Anthracycline chemotherapy [Count of Participants; unit: Participants] | 5
Prior therapy in any setting - Taxane chemotherapy [Count of Participants; unit: Participants] | 20
Prior therapy in any setting - Trastuzumab [Count of Participants; unit: Participants] | 20
Prior therapy in any setting - Pertuzumab [Count of Participants; unit: Participants] | 20
Prior therapy in any setting - T-DM1 [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: The number and type of DLTs as defined in the protocol that occur during the first 21 days of treatment and all maximum grade of all treatment-related adverse events using CTCAE v4.0 will be used to identify a safe and tolerable dose
Time Frame: 21 days
Population: The analysis population is patients that were enrolled in the dose de-escalation (dose finding) stage.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab Combine With Trastuzumab Emtansine: --All patients received 200mg Pembro + 3.6mg/kg T-DM1
  * Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * Pembrolizumab will be administered prior to T-DM1 administration
  * Pembrolizumab will be given at a predetermine dose
  * T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  * T-DM1 will be given at a predetermine dose
  T-DM1: -T-DM1 will be administered intravenousely in clinic on day 1 of each 3-week cycle
  Pembrolizumab: -Pembrolizumab will be administered intravenousely in clinic on day 1 of each 3-week cycle
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the percentage of patients with complete or partial response evaluated by RECIST 1.1. Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: All participants who have received at least one dose of study medication at the recommended phase 2 dose and had measurable disease were assessed for objective response rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
percentage of participants | 20 [5.7 to 43.7]

3. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival, estimated via Kaplan-Meier method, is defined as the time from study registration to radiographic evidence of disease progression or death due to any cause, whichever occurred first. Progression is measured using RECIST 1.1 criteria, defined as at least a 20% increase in size in target lesion and/or unequivocal progression of non-target lesions and/or appearance of new lesions. Patients alive without disease progression are censored at the date of last disease evaluation.
Time Frame: 2 years
Population: All participants who have received at least one dose of study medication at the recommended phase 2 dose were assessed for PFS
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
month | 9.6 [2.8 to 16]

4. Secondary Outcome: Duration Of Response
Description: The duration of response, estimated via Kaplan-Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Time Frame: 2 years
Population: All participants who have received at least one dose of study medication at the recommended phase 2 dose and had measurable disease were assessed for duration of response
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
month | 10.1 [3.1 to NA] — Upper limit for the 95% Confidence Interval could not be calculated due to an insufficient number of participants with events

5. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate will be determined by looking at the number of subjects who have either a complete response, partial response, or stable disease for greater than or equal to 18 weeks, per RECIST 1.1
Time Frame: 18 weeks
Population: All participants who have received at least one dose of study medication at the recommended phase 2 dose and had measurable disease were assessed for disease control rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
percentage of participants | 60 [36 to 80.9]

6. Secondary Outcome: Overall Survival Rate
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: 5 years
Population: All participants who have received at least one dose of study medication at the recommended phase 2 dose will be assessed for overall survival
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
Number analyzed (Participants) | 20
month | NA [11.2 to NA] — Median and upper limit for the 95% Confidence Interval could not be calculated due to an insufficient number of participants with events. The 50% survival probability was never reached due to small number of events. If a Kaplan-Meier curve is drawn, the curve will be above the 50% OS probability line. So no estimation could be made for median and the upper limit of confidence interval.

ADVERSE EVENTS:
Time Frame: AE data were collected every cycle from the time of the first dose of the study treatment, through the end of the treatment. Vital status was followed even after patients were off treatment. All-Cause Mortality was assessed up to 5 years, and all adverse events were collected up to 44 months.
Arm/Group | Pembrolizumab Combine With Trastuzumab Emtansine
All-Cause Mortality (participants affected / at risk) | 7/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Combine With Trastuzumab Emtansine (N=20)
Anemia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Hematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Combine With Trastuzumab Emtansine (N=20)
Anemia (Blood and lymphatic system disorders) | 5
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Heart failure (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 16
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 5
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 2
Bladder infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 8
Creatinine increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03032107/Prot_SAP_000.pdf